CLINICAL TRIAL: NCT06009848
Title: An Open ,Single Arm, Prospective, Phase II Clinical Study on the First-line Treatment of Recurrent or Metastatic Muscle Invasive Bladder Cancer With Cadonilimab(AK104) Plus Nab-Paclitaxel
Brief Title: Cadonilimab Plus Nab-Paclitaxel for Recurrent or Metastatic Muscle Invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-MIBC
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Bladder Cancer
Keywords: Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab (AK104) combined with Nab -Paclitaxel (Experimental): Cadonilimab (10 mg/kg, administered on the first day of each cycle, Q3W, until there is no clinical benefit)+Nab-Paclitaxel(200 mg/m2, Q3W, 6cycles), every 3 weeks (21 days) is a treatment cycle
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab (10 mg/kg, administered on the first day of each cycle, Q3W, until there is no clinical benefit)+Nab-Paclitaxel(200 mg/m2, Q3W ,6 cycles), every 3 weeks (21 days) is a treatment cycle.
  Other Names: AK104

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Cadonilimab(AK104) combined with Nab -Paclitaxel as first line therapy for recurrent or metastatic muscle invasive bladder. Eligible participants will receive AK104 (up to 24 months) plus Nab-Paclitaxel (for 6 cycles) until radiologic disease progression, unacceptable toxicity, or withdrawal from the study, whichever occurred first. The primary endpoint is objective response rate.

DETAILED DESCRIPTION:
Cadonilimab(AK104) is a first-in-class bispecific, humanized IgG1 antibody targeting PD-1 and CTLA-4, which has the potential to boost immune surveillance in tumors. The goal of this clinical phase II trial is to evaluate the efficacy and safety of AK104 combined with Nab-Paclitaxel as first line therapy for recurrent or metastatic muscle invasive bladder.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form before joining the group.
2. Age>18 years old.
3. Patients with advanced metastatic bladder cancer confirmed histologically or pathologically.
4. Have not received systemic treatment.
5. Have measurable lesions (according to RECIST 1.1 standard, non lymph node lesions have a CT scan length of ≥ 10 mm, and lymph node lesions have a CT scan short diameter of ≥ 15 mm).
6. ECOG PS score: 0-1.
7. The expected survival period is greater than 12 weeks.
8. The functions of important organs meet the following requirements (excluding the use of any blood components and cell growth factors within 14 days):

(1) Blood routine: Neutrophils ≥ 1.5 × 10^9/L;Platelet count ≥ 100 × 10^9/L;Hemoglobin ≥ 90g/L.

(2) Liver and kidney function:Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal value (ULN) or creatinine clearance rate ≥ 50 ml/min (Cockcroft Fault formula);Liver function: Aspartate aminotransferase (AST) ≤ 2.5 x ULN, alanine liver aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastasis; ALT and AST<5 x ULN in liver metastasis subjects.;Total serum bilirubin (TBIL) ≤ 1.5 x ULN (excluding Gilbert syndrome where TBIL<3.0 mg/dL);Urinary protein<2+;If the urine protein is ≥ 2+, the 24-hour urine protein quantitative display must be ≤ 1g.

9. Normal coagulation function, no active bleeding or thrombosis disease

1. International standardized ratio INR ≤ 1.5 × ULN;
2. Partial thromboplastin time APTT ≤ 1.5 × ULN;
3. Prothrombin time PT ≤ 1.5 × ULN. 10. Non surgical sterilization or reproductive age female patients are required to use a medically approved contraceptive method (such as an intrauterine device, contraceptive pill, or condom) during the study treatment period and within 3 months after the end of the study treatment period. Non surgically sterilized female patients of childbearing age must have a negative serum or urine HCG test within 7 days before enrollment in the study. And it must be non lactating.

11. The subjects voluntarily joined this study with good compliance, safety, and survival follow-up.

Exclusion Criteria:

1. The subject has previously or simultaneously suffered from other malignant tumors (excluding cured skin basal cell carcinoma and cervical carcinoma in situ).
2. The subject is known to have previous allergies to macromolecular protein formulations or known to be allergic to the drug components used.
3. The subject has any active autoimmune disease or a history of autoimmune disease (For example, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, decreased thyroid function, who have undergone thyroid surgery in the past cannot be included. subjects with vitiligo or complete remission of childhood asthma, who do not require any intervention in adulthood, can be included. subjects who require bronchodilators for medical intervention) Asthma cannot be included).
4. The subject is currently using immunosuppressive agents or systemic or absorbable local hormone therapy to achieve immunosuppressive effects (dosage>10mg/day of prednisone or other therapeutic hormones), and continues to use them within 2 weeks before enrollment.
5. Ascites or pleural effusion with clinical symptoms require therapeutic puncture or drainage.
6. Patients with clinically uncontrollable cardiac symptoms or diseases, such as: (1) NYHA grade 2 or above heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias that require treatment or intervention.
7. The subject has an active infection or an unexplained fever>38.5 degrees Celsius during the screening period or before the first administration (according to the researcher's judgment, the subject's fever caused by the tumor can be included in the group).
8. Patients with past and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, and severe impairment of lung function with objective evidence.
9. Subjects have congenital or acquired immune deficiency, such as HIV infected persons, or active hepatitis (transaminase does not meet the inclusion criteria, hepatitis B reference: HBV DNA ≥ 1000 IU/ml. hepatitis C reference: HCV RNA ≥ 1000 IU/ml). Chronic hepatitis B virus carriers with HBV DNA<2000 IU/ml must receive antiviral treatment simultaneously during the trial period before they can be enrolled.
10. Live vaccines may be administered less than 4 weeks before the study medication or during the study period.
11. The subject is known to have a history of psychotropic substance abuse, alcoholism, or drug abuse.
12. Accepted Chinese herbal medicine or traditional Chinese patent medicines and simple preparations with anti-tumor indications within 2 weeks before the first administration.
13. The researcher believes that it should be excluded from this study. For example, based on the researcher's judgment, the subject may have other factors that may cause the study to be terminated midway, such as other serious diseases (including mental illness) requiring concurrent treatment, serious laboratory test abnormalities, accompanied by family or social factors, which may affect the safety of the subject, or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | The last subject completes at least 24 weeks of follow-up (or disease progression)
  The proportion of patients whose tumor volume is reduced to 30% and can be maintained for more than 4 weeks,Based on RECIST v1.1.

SECONDARY OUTCOMES:
Overall Survival(OS) | 24 months
  The time from the patient receiving treatment to the death of the patient for any reason,OS evaluated according to RECIST v1.1.
Progression-free Survival(PFS) | The last subject completes at least 24 weeks of follow-up (or disease progression)
  The time from the beginning of the patient's treatment to the disease progression or death for any reason.Based on RECIST v1.1.
Duration of Response(DOR) | The last subject completes at least 24 weeks of follow-up (or disease progression)
  Duration of response (DOR) as assessed by the investigator according to RECIST v1.1.
Adverse events(AEs） | 24 months
  Include Treatment emerge adverse events, treatment related adverse events and serious adverse events,AEs evaluated according to NCI-CTCAE v5.0 and irAE.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China